CLINICAL TRIAL: NCT00599963
Title: Paricalcitol for the Treatment of Immunoglobulin A Nephropathy - A Randomized Cross-Over Study
Brief Title: Paricalcitol for the Treatment of Immunoglobulin A Nephropathy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding problem.
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Dr. SZETO, Cheuk Chun, The Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2007.409-T; CRE-2007.409-T
Record Dates: First submitted 2008-01-02; First posted 2008-01-24 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2009-01

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): paricalcitol 1 mg/day for 12 weeks, followed by a washout period of 4 weeks, then crossed over to no treatment for another 12 weeks
  Interventions: Drug: paricalcitol
- 2 (Active Comparator): no treatment for 12 weeks, followed by a washout period of 4 weeks, then crossed over to paricalcitol for another 12 weeks
  Interventions: Drug: paricalcitol

INTERVENTIONS:
Drug: paricalcitol — paricalcitol 1 mg/day

SUMMARY:
Immunoglobulin A (IgA) nephropathy is the common type of primary glomerulonephritis in the world. A wealth of literature suggests that vitamin D and its analogs have profound effects on immune system function and glomerular mesangial cell proliferation. However, calcitriol, the standard form of vitamin D, carries a substantial risk of hypercalcemia. Recently, paricalcitol (19-nor-1,25-dihydroxyvitamin D2) was approved for the treatment of secondary hyperparathyroidism in chronic renal failure, and the incidence of hypercalcemia is much lower than calcitriol. Therefore, the investigators plan to conduct a randomized cross-over study to evaluate the efficacy of paricalcitol in the treatment of IgA nephropathy. Thirty patients with biopsy-proven IgA nephropathy will be recruited. They will be randomized to paricalcitol for 12 weeks or no treatment, followed by cross over to the other arm after a washout period. Proteinuria, renal function, serum and urinary inflammatory markers will be monitored. This study will explore the potential anti-proteinuric and anti-inflammatory effects of paricalcitol in the treatment of IgA nephropathy, which has no specific treatment at present.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* biopsy-confirmed IgA nephropathy
* proteinuria > 1 g/day (or proteinuria > 1 g/g-Cr) in 3 consecutive samples within 12 weeks despite ACE inhibitor or angiotensin receptor blocker treatment (e.g. ramipril 5 mg daily, lisinopril 10 mg daily, or valsartan 80 mg daily) for at least 3 months
* estimated glomerular filtration rate > 60 ml/min/1.73m2
* corrected serum calcium level > or = 2.45 mmol/l
* willingness to give written consent and comply with the study protocol

Exclusion Criteria:

* Pregnancy, lactating or childbearing potential without effective method of birth control
* Severe gastrointestinal disorders that interfere with their ability to receive or absorb oral medication
* History of malignancy, including leukemia and lymphoma within the past 2 years
* Systemic infection requiring therapy at study entry
* Any other severe coexisting disease such as, but not limited to, chronic liver disease, myocardial infarction, cerebrovascular accident, malignant hypertension
* History of drug or alcohol abuse within past 2 years
* Participation in any previous trial on paricalcitol
* Patients receiving treatment of vitamin D and/or its analogue for other medical reasons within the past 3 months
* Patients receiving treatment of corticosteroid
* On other investigational drugs within last 30 days
* History of a psychological illness or condition such as to interfere with the patient's ability to understand the requirement of the study
* History of non-compliance
* Known history of sensitivity or allergy to paricalcitol or other vitamin D analogs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
change in the degree of proteinuria | 12 weeks

SECONDARY OUTCOMES:
rate of decline of estimated GFR (as determined by the least square method) and change in other serum inflammatory markers | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cheuk Chun Szeto, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Medicine & Therapeutics, Prince of Wales Hospital, Shatin, Hong Kong